CLINICAL TRIAL: NCT03362905
Title: Lidocaine for Pain Control During Intrauterine Device Insertion: A Randomized Clinical Trial
Brief Title: Lidocaine for Pain Control During Intrauterine Device Insertion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hadeer Abd-El Shafy Fouad, Resident physician, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lidocaine in IUD pain
Record Dates: First submitted 2017-11-30; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: IUD Insertion Complication
Keywords: Lidocaine; Dosage forms; Pain scores
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: This study will include 123 patients who are candidates for IUD contraception. The aim of the study will be explained to all patients and an informed written consent will be taken. After recruitment, patients will be randomized to the 3 study arms using computer generated randomization sheet using MedCalcc version 13 to receive any of: lidocaine spray, cream and injection
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine spray Arm (Experimental): This arm will receive lidocaine spray (Lidocaine topical aerosol ®, 10%, Arab drug co., Egypt) with dose four puffs (50 ml, 10 mg/puff) will be applied to the cervical canal and cervix.
  Interventions: Drug: Lidocaine topical
- Lidocaine cream Arm (Active Comparator): This arm will receive topical cream (Pridocaine ®, Global Napi, Egypt) with a dose of 2g lidocaine cream will be applied to the cervix via cotton swab.
  Interventions: Drug: Lidocaine topical
- Lidocaine injection Arm (Active Comparator): This arm will receive lidocaine injection (Debocaine®, 2%, Sigma-Tec, Egypt) with a dose of 80-200 mg equivalent to 10 ml lidocaine (20 mg/ml) is injected at four and eight o'clock of the cervico-vaginal junction, and 2 ml to the area to be grasped with the tenaculum for paracervical block.
  Interventions: Drug: Lidocaine topical

INTERVENTIONS:
Drug: Lidocaine topical — Local anesthetic for reduction of IUD associated pain

SUMMARY:
Despite being the most common method of contraception, the use of intrauterine devices (IUDs) is limited by the associated pain during insertion. Many pharmacologic interventions had been studied for their efficacy to reduce IUD insertion pain, of them, lidocaine was found to be superior over NSAIDs or other local anesthetics. This work aims at comparing the safety and efficacy of different lidocaine formulations to optimize selection in reduction of IUD associated pain.

ELIGIBILITY:
Inclusion Criteria:

1. Multiparous women.
2. Over 18 years of age and eligible for IUD insertion.
3. Application of IUD will be done in postmenstrual period.

Exclusion Criteria:

Null parity. 2. History of failed intrauterine device insertion (uterine perforation, acute expulsion).

3. Copper allergy. 4. Uterine anomaly. 5. Post-partum endometritis or septic abortion in the past three months. 6. Untreated cervicitis/vaginitis, including bacterial vaginosis. 7. Immunosuppression. 8. History of lidocaine ,prilocaine allergy. 9. Analgesic or anxiolytic use within the last 24 hours before the procedure. 10. Wilson's disease. 11. Suspicion of pregnancy. 12. Untreated abnormal uterine bleeding.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Estimated)
Dates: Start 2017-12-03 (Estimated); Primary Completion 2018-12-05 (Estimated); Study Completion 2019-01-10 (Estimated)

PRIMARY OUTCOMES:
Pain scores assessed by 10-point VAS scale | 1 year
  VAS scores will be assessed on at three different points; baseline after application of speculum and analgesic administration, after grasping cervix with tenaculum, then following hysterometry and IUD insertion.

SECONDARY OUTCOMES:
Patient satisfaction to IUD insertion | 1 year
  Satisfaction will be assessed post-procedure using patient directed survey

REFERENCES:
- [Background] Aksoy H, Aksoy U, Ozyurt S, Acmaz G, Babayigit M. Lidocaine 10% spray to the cervix reduces pain during intrauterine device insertion: a double-blind randomised controlled trial. J Fam Plann Reprod Health Care. 2016 Apr;42(2):83-7. doi: 10.1136/jfprhc-2014-100917. Epub 2015 Mar 10. PMID 25759418
- [Background] Buhling KJ, Hauck B, Dermout S, Ardaens K, Marions L. Understanding the barriers and myths limiting the use of intrauterine contraception in nulliparous women: results of a survey of European/Canadian healthcare providers. Eur J Obstet Gynecol Reprod Biol. 2014 Dec;183:146-54. doi: 10.1016/j.ejogrb.2014.10.020. Epub 2014 Oct 30. PMID 25461369
- [Background] Lopez LM, Bernholc A, Zeng Y, Allen RH, Bartz D, O'Brien PA, Hubacher D. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2015 Jul 29;2015(7):CD007373. doi: 10.1002/14651858.CD007373.pub3. PMID 26222246
- [Background] Gemzell-Danielsson K, Mansour D, Fiala C, Kaunitz AM, Bahamondes L. Management of pain associated with the insertion of intrauterine contraceptives. Hum Reprod Update. 2013 Jul-Aug;19(4):419-27. doi: 10.1093/humupd/dmt022. Epub 2013 May 12. PMID 23670222
- [Background] Bahamondes L, Mansour D, Fiala C, Kaunitz AM, Gemzell-Danielsson K. Practical advice for avoidance of pain associated with insertion of intrauterine contraceptives. J Fam Plann Reprod Health Care. 2014 Jan;40(1):54-60. doi: 10.1136/jfprhc-2013-100636. Epub 2013 Sep 27. PMID 24076534
- [Background] Akers AY, Steinway C, Sonalkar S, Perriera LK, Schreiber C, Harding J, Garcia-Espana JF. Reducing Pain During Intrauterine Device Insertion: A Randomized Controlled Trial in Adolescents and Young Women. Obstet Gynecol. 2017 Oct;130(4):795-802. doi: 10.1097/AOG.0000000000002242. PMID 28885425
- [Background] Tavakolian S, Doulabi MA, Baghban AA, Mortazavi A, Ghorbani M. Lidocaine-Prilocaine Cream as Analgesia for IUD Insertion: A Prospective, Randomized, Controlled, Triple Blinded Study. Glob J Health Sci. 2015 Jan 27;7(4):399-404. doi: 10.5539/gjhs.v7n4p399. PMID 25946948
- [Background] Golzari SE, Soleimanpour H, Mahmoodpoor A, Safari S, Ala A. Lidocaine and pain management in the emergency department: a review article. Anesth Pain Med. 2014 Feb 15;4(1):e15444. doi: 10.5812/aapm.15444. eCollection 2014 Feb. PMID 24660158
- [Background] Mody SK, Kiley J, Rademaker A, Gawron L, Stika C, Hammond C. Pain control for intrauterine device insertion: a randomized trial of 1% lidocaine paracervical block. Contraception. 2012 Dec;86(6):704-9. doi: 10.1016/j.contraception.2012.06.004. Epub 2012 Jul 6. PMID 22770792